CLINICAL TRIAL: NCT00988767
Title: Specific Vaccine Therapy in Chronic Hepatitis B Using a Naked DNA: Phase I Study Using a GMO
Brief Title: Safety and Immunogenicity of a Naked DNA-based Vaccine Therapy in Patients With Chronic Hepatitis B
Acronym: RBM99026
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INSERM RBM99.026
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Last update posted 2025-09-26 (Actual); Status verified 2009-10

CONDITIONS: Chronic Hepatitis B
Keywords: Hepatitis B; DNA vaccine; immunotherapy
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — Vaccines, DNA

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- intramuscular injections (Experimental): Patients received 4 injections of DNA vaccine at M0, M2, M4 and M10
  Interventions: Biological: DNA vaccine

INTERVENTIONS:
Biological: DNA vaccine — patients received 1ml of DNA vaccine (1mg/ml) at Months 0,2,4,10
  Other Names: pCMV-S2.S DNA

SUMMARY:
The purpose of this study was to investigate whether HBV-DNA vaccination is safe and could restore immune responses in patients with chronic hepatitis B non responder to available therapies.

DETAILED DESCRIPTION:
* Despite the availability of effective hepatitis B vaccines for many years, over 370 million people remain persistently infected with hepatitis B virus (HBV). Persistent infection is associated with chronic liver disease that can lead to the development of cirrhosis and hepatocellular carcinoma in some patients. Viral persistence is thought to be related to poor HBV-specific immune responses.
* Interferon (IFN)-alpha treatment significantly decreases HBV replication in only one third of patients with hepatitis B e antigen (HBeAg)-positive chronic active hepatitis B. Nucleoside analogues, such as lamivudine and adefovir dipivoxil, inhibit HBV replication and improve histological signs of liver disease,but their use is limited by the risk of relapse after treatment discontinuation and the emergence of drug-resistant viral variants.
* Patients with acute self-limited hepatitis B display detectable polyclonal and multispecific cytotoxic T lymphocyte and T helper (Th) responses to viral antigens,whereas these responses are weak or absent in chronic HBV carriers.
* Increasing the strength of HBV-specific T-cell responses to the levels found in patients recovering from infection is therefore a goal in the treatment of patients with chronic hepatitis.
* Immunization with a nucleic acid vaccine (DNA vaccine) usually elicits antibody responses and T lymphocytes with a Th1 cytokine profile. In animal models of chronic hepatitis B infection, including nonhuman primates, intramuscular injection of a plasmid encoding HBV envelope proteins induces rapid, strong, and sustained humoral and cell-mediated immune responses. Clinical trials of DNA vaccines for hepatitis B conducted in healthy adult volunteers using a plasmid encoding hepatitis B surface antigen and the gene gun as a delivery system showed good tolerance.
* We carried out a phase I trial of a HBV DNA vaccine in patients with chronic active viral hepatitis, aiming to restore HBV-specific immune responses and to assess safety regarding liver disease.

ELIGIBILITY:
Inclusion Criteria:

* chronic HBV carriers
* biopsy proven chronic hepatitis
* active HBV replication for > 6 months
* non responding to Interferon-alpha or lamivudine treatment

Exclusion Criteria:

* co-infection with HIV, HCV, delta hepatitis virus
* alcohol consumption> 40g/day
* decompensated liver disease
* HLA DR2

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2001-02; Primary Completion 2003-11 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability (local and general) of the DNA vaccine injections | every Months from month 0 to month 12 and then M15, M18, M21 and M22

SECONDARY OUTCOMES:
Immunological responses | before DNA injection (M0), after DNA injection and during follow-up (M1, M3, M5, M10, M11, M15)

CONTACTS AND LOCATIONS:
Overall Officials: Helene FONTAINE, MD, Principal Investigator — Assistance Publique des Hopitaux de paris, AP-HP
Locations (1):
- Service d'Hepatologie, Hopital Necker Enfants Malades, Paris, France

REFERENCES:
- [Background] Mancini-Bourgine M, Fontaine H, Scott-Algara D, Pol S, Brechot C, Michel ML. Induction or expansion of T-cell responses by a hepatitis B DNA vaccine administered to chronic HBV carriers. Hepatology. 2004 Oct;40(4):874-82. doi: 10.1002/hep.20408. PMID 15382173
- [Background] Mancini-Bourgine M, Fontaine H, Brechot C, Pol S, Michel ML. Immunogenicity of a hepatitis B DNA vaccine administered to chronic HBV carriers. Vaccine. 2006 May 22;24(21):4482-9. doi: 10.1016/j.vaccine.2005.08.013. Epub 2005 Aug 18. PMID 16310901
- [Derived] Scott-Algara D, Mancini-Bourgine M, Fontaine H, Pol S, Michel ML. Changes to the natural killer cell repertoire after therapeutic hepatitis B DNA vaccination. PLoS One. 2010 Jan 18;5(1):e8761. doi: 10.1371/journal.pone.0008761. PMID 20090916